CLINICAL TRIAL: NCT05249270
Title: Online Parent-Report Evaluation of the Effects of Processed Music
Status: Terminated | Type: Observational
Why Stopped: Inadequate resources ot complete data collection during COVID pandemic
Sponsor: Indiana University (Other)
Collaborators: Children's Therapy of Woodinville (Unknown)
Responsible Party: Principal Investigator, Jacek Kolacz, Assistant Research Scientist, Indiana University
Other Study IDs: 1912463776
Record Dates: First submitted 2021-03-19; First posted 2022-02-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Sensory Disorders; Sensory Processing Disorder; Autism Spectrum Disorder; Eating Disorders; Gastro-Intestinal Disorder; Swallowing Disorder; Anxiety
MeSH Terms: conditions — Sensation Disorders; Autism Spectrum Disorder; Feeding and Eating Disorders; Digestive System Diseases; Deglutition Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Safe and Sound Protocol Participants: Parents of children receiving the Safe and Sound Protocol (a clinical auditory therapy provided outside of the study) will complete questionnaires to assess sensory behaviors prior to therapy initiation (baseline), 1 week after therapy conclusion, and 4 weeks after therapy conclusion. The SSP typically consists of 1 hour of listening per day, for 5 consecutive days. If modifications of the typical dosage are implemented due to client needs, they will be documented by parents in the 1 week post therapy questionnaire.

SUMMARY:
The study aims to examine effectiveness of the Safe and Sound Protocol (SSP) on sensory, digestive, and eating behaviors in children currently receiving therapy.

DETAILED DESCRIPTION:
The SSP consists of listening to a computer altered sequence of vocal music that has been processed to "exercise" the neural regulation of the middle ear muscles. Low and high frequencies are dynamically filtered and presented monaurally to both ears. The intervention stimuli are delivered through headphones or speakers. The protocol consists of 60 minutes of listening on five sequential days and is delivered via a music player device in a quiet room without major distractors.

For this study, parents or legal guardians of children already enrolled to complete the SSP intervention at Children's Therapy of Woodinville will complete a series of surveys. The SSP is used as a component of therapy across multiple diagnostic categories including autism spectrum disorders and sensory processing disorder. No specific diagnoses will be targeted in this design. Parents will be recruited for the study if their child is already enrolled to receive the therapy. Participating parents will be asked to complete online questionnaires using a survey link at three intervals: before the start of therapy, one week after completion, and 1 month after completion.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of child who is receiving the Safe and Sound Protocol at Children's Therapy of Woodinville (in Woodinville, WA)
* Parent must be 18 years or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parents or legal guardians of children who are receiving the Safe and Sound Protocol at Children's Therapy of Woodinville (in Woodinville, WA)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Sensory sensitivities | Change from baseline to 1 and 4 week post assessment
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

SECONDARY OUTCOMES:
Selective eating | Change from baseline to 1 and 4 week post assessment
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)
Ingestive problems | Change from baseline to 1 and 4 week post assessment
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)
Digestive problems | Change from baseline to 1 and 4 week post assessment
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Therapy of Woodinville, Woodinville, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porges SW, Bazhenova OV, Bal E, Carlson N, Sorokin Y, Heilman KJ, Cook EH, Lewis GF. Reducing auditory hypersensitivities in autistic spectrum disorder: preliminary findings evaluating the listening project protocol. Front Pediatr. 2014 Aug 1;2:80. doi: 10.3389/fped.2014.00080. eCollection 2014. PMID 25136545
- [Background] Porges SW, Macellaio M, Stanfill SD, McCue K, Lewis GF, Harden ER, Handelman M, Denver J, Bazhenova OV, Heilman KJ. Respiratory sinus arrhythmia and auditory processing in autism: modifiable deficits of an integrated social engagement system? Int J Psychophysiol. 2013 Jun;88(3):261-70. doi: 10.1016/j.ijpsycho.2012.11.009. Epub 2012 Nov 29. PMID 23201146